CLINICAL TRIAL: NCT05258292
Title: Glycemic Variations During the Menstrual Cycle in Women With Type 1 Diabetes: the GLYMETY Study
Brief Title: Glycemic Variations During the Menstrual Cycle in Women With Type 1 Diabetes
Acronym: GLYMETY
Status: Recruiting | Type: Observational
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Full professor, Institut de Recherches Cliniques de Montreal
Other Study IDs: 2022-1165
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Type1diabetes
Keywords: Menstrual cycle; Continuous glucose monitoring; Insulin dose; Physical activity; Food intake
MeSH Terms: conditions — Motor Activity | interventions — Continuous Glucose Monitoring; Insulin; Menstrual Cycle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with type 1 diabetes
  Interventions: Device: Continuous glucose monitoring; Drug: Insulin; Other: Premenstrual symptoms; Other: Ovulation kits; Device: Fitbit Inspire 2; Other: Keenoa; Other: Menstrual cycle

INTERVENTIONS:
Device: Continuous glucose monitoring — Glucose levels will be measured using continuous glucose monitoring
Drug: Insulin — Insulin doses will be retrieved from insulin pump reports (for insulin pump users) or journals for (for multiple daily injections users)
Other: Premenstrual symptoms — Premenstrual symptoms will be assessed using the Premenstrual symptoms screening tool
Other: Ovulation kits — Ovulation testing will be done using ovulation kits
Device: Fitbit Inspire 2 — Physical activity will be assessed using the Fitbit Inspire 2
Other: Keenoa — Food intake will be assessed using the Keenoa phone application
Other: Menstrual cycle — The application My Calendar will be used to record information on the menstrual cycle

SUMMARY:
In clinical practice, women living with type 1 diabetes frequently report that insulin requirements change across the menstrual cycle. Consequently, glycemic fluctuations are observed. This phenomenon could be explained by a decrease in insulin sensitivity during the second half of the menstrual cycle (luteal phase).

Overall, despite an important proportion of women reporting glycemic and/or insulin variations across the menstrual cycle, studies to date have involved small sample sizes, and have had inconsistent results. The objective of this study will be to study glycemic fluctuations across the menstrual cycle using CGM data, alongside insulin data, in a large sample of women.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18 to 50 living in Canada.
2. Clinical diagnosis of type 1 diabetes or latent autoimmune diabetes in adults (LADA) for at least one year.
3. Using insulin pump therapy, multiple daily injections or automated insulin delivery systems for at least 3 months.
4. Using a continuous glucose monitoring (CGM) system.
5. Having at least one menses in the last 40 days.
6. Accepting to share CGM data with the research team and if applicable insulin pump data.This access will be limited to the study period.
7. Having a smartphone or tablet to follow menstrual cycles.
8. Stable weight (less than 5% variation in the last 3 months).

Exclusion Criteria:

1. Using a hormonal contraception method that eliminates menses (Depo Provera, progestin intrauterine device, extented-cycle regimen with birth control pill)
2. Using regular insulin (Entuzity U500, Novolin ge Toronto or Humulin R).
3. Clinically significant nephropathy (eGFR < 30 ml/min/1.73m2, planned or on dialysis) or neuropathy (e.g., known uncontrolled gastroparesis) as judged by the investigator.
4. Recent (< 6 months) acute macrovascular event (e.g., acute coronary syndrome or cardiac surgery).
5. Anticipated therapeutic change (including change of insulin type and/or type of CGM sensor, insulin pump or AID (automated insulin device) system) between admission and end of the study.
6. Anticipated change in contraception method or plan to begin or stop a contraceptive method.
7. Anticipated need to use acetaminophen during the study period at a dose above 1g every 6 hours.
8. Pregnancy (ongoing or current attempt to become pregnant)
9. Breastfeeding
10. Uncontrolled thyroid disease (TSH should be in target range and treatment stable for at least 6 weeks).
11. Severe hypoglycemic episode within two weeks of screening
12. Severe hyperglycemic episodes requiring hospitalization in the last 3 months.
13. Current use of glucocorticoid medication (except low stable dose and inhaled steroids and stable adrenal insufficiency treatment e.g., Cortef®)
14. Agents affecting gastric emptying (Motilium®, Victoza®, Ozempic®, Trulicity®, Byetta® and Symlin®) as well as oral anti-diabetic agents (Metformin, Prandase®, DPP-4 inhibitors) unless at a stable dose for 3 months and without anticipated change during the study.
15. Current use of SGLT-2 inhibitors unless at a stable dose for at least 3 months, without anticipated change during the study and appropriate ketone testing is performed.
16. Other serious medical illnesses which likely interfere with study participation or with the ability to complete the study by the judgment of the investigator.
17. Anticipation of a significant change in exercise or diet regimen between admission and end of the study (i.e., starting or stopping an organized sport; planned significant diet change).
18. Anticipated radiologic examination incompatible with CGM wear for more than 10 days between admission and end of the study (e.g., repeated MRI).
19. In the opinion of the investigator, a participant who is unable or unwilling to complete the study.
20. If taking medication for hypothyroidism, no change of dose (Levothyroxin) in the last 6 weeks.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 18 to 50 living with type 1 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Mean glucose levels during the early follicular phase | Day 1 to 5 of the menstrual cycle
Mean glucose levels during the mid-late follicular phase | Day 6 until 2 days prior to ovulation
Mean glucose levels during the periovulation phase | Ovulation plus/minus 1 day
Mean glucose levels during the early luteal phase | Day 2 to 4 after ovulation
Mean glucose levels during the mid-luteal phase | Day 5 to 9 after ovulation
Mean glucose levels during the late luteal phase | Day 10 after ovulation until the first day of the next menstrual cycle

SECONDARY OUTCOMES:
Percentage of time of glucose levels between 3.9 and 7.8 mmol/L | Day 1 to 5 of the menstrual cycle
Percentage of time of glucose levels between 3.9 and 7.8 mmol/L | Day 6 until 2 days prior to ovulation
Percentage of time of glucose levels between 3.9 and 7.8 mmol/L | Ovulation plus/minus 1 day
Percentage of time of glucose levels between 3.9 and 7.8 mmol/L | Day 2 to 4 after ovulation
Percentage of time of glucose levels between 3.9 and 7.8 mmol/L | Day 5 to 9 after ovulation
Percentage of time of glucose levels between 3.9 and 7.8 mmol/L | Day 10 after ovulation until the first day of the next menstrual cycle
Percentage of time of glucose levels between 3.9 and 10.0 mmol/L | Day 1 to 5 of the menstrual cycle
Percentage of time of glucose levels between 3.9 and 10.0 mmol/L | Day 6 until 2 days prior to ovulation
Percentage of time of glucose levels between 3.9 and 10.0 mmol/L | Ovulation plus/minus 1 day
Percentage of time of glucose levels between 3.9 and 10.0 mmol/L | Day 2 to 4 after ovulation
Percentage of time of glucose levels between 3.9 and 10.0 mmol/L | Day 5 to 9 after ovulation
Percentage of time of glucose levels between 3.9 and 10.0 mmol/L | Day 10 after ovulation until the first day of the next menstrual cycle
Percentage of time of glucose levels below 3.9 mmol/L | Day 1 to 5 of the menstrual cycle
Percentage of time of glucose levels below 3.9 mmol/L | Day 6 until 2 days prior to ovulation
Percentage of time of glucose levels below 3.9 mmol/L | Ovulation plus/minus 1 day
Percentage of time of glucose levels below 3.9 mmol/L | Day 2 to 4 after ovulation
Percentage of time of glucose levels below 3.9 mmol/L | Day 5 to 9 after ovulation
Percentage of time of glucose levels below 3.9 mmol/L | Day 10 after ovulation until the first day of the next menstrual cycle
Percentage of time of glucose levels below 3.0 mmol/L | Day 1 to 5 of the menstrual cycle
Percentage of time of glucose levels below 3.0 mmol/L | Day 6 until 2 days prior to ovulation
Percentage of time of glucose levels below 3.0 mmol/L | Ovulation plus/minus 1 day
Percentage of time of glucose levels below 3.0 mmol/L | Day 2 to 4 after ovulation
Percentage of time of glucose levels below 3.0 mmol/L | Day 5 to 9 after ovulation
Percentage of time of glucose levels below 3.0 mmol/L | Day 10 after ovulation until the first day of the next menstrual cycle
Percentage of time of glucose levels above 10.0 mmol/L | Day 1 to 5 of the menstrual cycle
Percentage of time of glucose levels above 10.0 mmol/L | Day 6 until 2 days prior to ovulation
Percentage of time of glucose levels above 10.0 mmol/L | Ovulation plus/minus 1 day
Percentage of time of glucose levels above 10.0 mmol/L | Day 2 to 4 after ovulation
Percentage of time of glucose levels above 10.0 mmol/L | Day 5 to 9 after ovulation
Percentage of time of glucose levels above 10.0 mmol/L | Day 10 after ovulation until the first day of the next menstrual cycle
Percentage of time of glucose levels above 13.9 mmol/L | Day 1 to 5 of the menstrual cycle
Percentage of time of glucose levels above 13.9 mmol/L | Day 6 until 2 days prior to ovulation
Percentage of time of glucose levels above 13.9 mmol/L | Ovulation plus/minus 1 day
Percentage of time of glucose levels above 13.9 mmol/L | Day 2 to 4 after ovulation
Percentage of time of glucose levels above 13.9 mmol/L | Day 5 to 9 after ovulation
Percentage of time of glucose levels above 13.9 mmol/L | Day 10 after ovulation until the first day of the next menstrual cycle
Standard deviation of glucose levels | Day 1 to 5 of the menstrual cycle
Standard deviation of glucose levels | Day 6 until 2 days prior to ovulation
Standard deviation of glucose levels | Ovulation plus/minus 1 day
Standard deviation of glucose levels | Day 2 to 4 after ovulation
Standard deviation of glucose levels | Day 5 to 9 after ovulation
Standard deviation of glucose levels | Day 10 after ovulation until the first day of the next menstrual cycle
Coefficient of variance of glucose levels | Day 1 to 5 of the menstrual cycle
Coefficient of variance of glucose levels | Day 6 until 2 days prior to ovulation
Coefficient of variance of glucose levels | Ovulation plus/minus 1 day
Coefficient of variance of glucose levels | Day 2 to 4 after ovulation
Coefficient of variance of glucose levels | Day 5 to 9 after ovulation
Coefficient of variance of glucose levels | Day 10 after ovulation until the first day of the next menstrual cycle
Low blood glucose index | Day 1 to 5 of the menstrual cycle
Low blood glucose index | Day 6 until 2 days prior to ovulation
Low blood glucose index | Ovulation plus/minus 1 day
Low blood glucose index | Day 2 to 4 after ovulation
Low blood glucose index | Day 5 to 9 after ovulation
Low blood glucose index | Day 10 after ovulation until the first day of the next menstrual cycle
High blood glucose index | Day 1 to 5 of the menstrual cycle
High blood glucose index | Day 6 until 2 days prior to ovulation
High blood glucose index | Ovulation plus/minus 1 day
High blood glucose index | Day 2 to 4 after ovulation
High blood glucose index | Day 5 to 9 after ovulation
High blood glucose index | Day 10 after ovulation until the first day of the next menstrual cycle
Standard deviation of insulin delivery | Day 1 to 5 of the menstrual cycle
Standard deviation of insulin delivery | Day 6 until 2 days prior to ovulation
Standard deviation of insulin delivery | Ovulation plus/minus 1 day
Standard deviation of insulin delivery | Day 2 to 4 after ovulation
Standard deviation of insulin delivery | Day 5 to 9 after ovulation
Standard deviation of insulin delivery | Day 10 after ovulation until the first day of the next menstrual cycle
Coefficient of variance of insulin delivery | Day 1 to 5 of the menstrual cycle
Coefficient of variance of insulin delivery | Day 6 until 2 days prior to ovulation
Coefficient of variance of insulin delivery | Ovulation plus/minus 1 day
Coefficient of variance of insulin delivery | Day 2 to 4 after ovulation
Coefficient of variance of insulin delivery | Day 5 to 9 after ovulation
Coefficient of variance of insulin delivery | Day 10 after ovulation until the first day of the next menstrual cycle
Total insulin delivery | Day 1 to 5 of the menstrual cycle
Total insulin delivery | Day 6 until 2 days prior to ovulation
Total insulin delivery | Ovulation plus/minus 1 day
Total insulin delivery | Day 2 to 4 after ovulation
Total insulin delivery | Day 5 to 9 after ovulation
Total insulin delivery | Day 10 after ovulation until the first day of the next menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No